CLINICAL TRIAL: NCT00213746
Title: Prediction of Left Ventricular Function Changes Using Low Dose Dobutamine Gated SPECT in Patients Referred for Viability Assessment: The DOGS (DObutamine Gated Spect)Study.
Brief Title: Evaluation of Myocardial Viability by Means of Low-dose Dobutamine Gated SPECT (the DOGS Study)
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Collaborators: Bristol-Myers Squibb (Industry); GE Healthcare (Industry); Fédération Française de Cardiologie (Other); Société Française de Cardiologie (Other); Société Française de Médecine Nucléaire (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2003/011/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Coronary Arteriosclerosis; Heart Failure, Congestive; Myocardial Infarction; Myocardial Ischemia; Myocardial Stunning
Keywords: Coronary Arteriosclerosis; Heart Failure, Congestive; Myocardial Infarction; Myocardial Revascularization; Tomography, Emission-Computed, Single-Photon; Dobutamine; Myocardial Stunning; Myocardial Hibernation
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure; Myocardial Infarction; Myocardial Ischemia; Myocardial Stunning

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Viability assessment remains a clinical challenge in patient with coronary artery disease and left ventricular dysfunction. Several imaging modalities are available for evaluating myocardial viability, based either on perfusion or on contractile reserve analysis. Briefly, perfusion analysis is highly sensitive and contractile reserve highly specific. A combined analysis of both perfusion and contractile reserve has been proposed to improve the diagnostic accuracy in patient referred for a revascularization procedure. However, the value of this combined analysis has not been validated in unselected patients referred for viability assessment.

The patients enrolled in the study will undergo a nitrate enhanced rest gated SPECT using a Tc-99m labeled tracer (sestamibi or tetrofosmine) followed by a second gated SPECT acquired during a low-dose dobutamine infusion (10 mcg/kg/mn). All patients will have a 6-month clinical and imaging follow-up, including physical examination and a nitrate enhanced rest gated SPECT using the same radiopharmaceutical. All treatments received during this 6-month period will be recorded, including medical therapy and coronary revascularization (angioplasty, stenting and CABG).

Finally, the value of baseline perfusion and contractile reserve analysis in predicting left ventricular ejection fraction changes at 6-month follow-up will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Documented coronary artery disease
* Left ventricular dysfunction (LVEF < 50%)
* Patients referred to the Nuclear Medicine department for myocardial viability assessment
* Sinus Rhythm
* Acceptance of a 6-month follow-up
* Signed informed consent

Exclusion Criteria:

* Recent acute coronary syndrome (< 21 days)
* Atrial Fibrillation or significant arrhythmias
* Implanted pacemaker
* Contra indication to dobutamine
* Non ischaemic cardiomyopathy
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists with patients with documented coronary artery disease and left ventricular dysfunction (LVEF < 50%)referred to aNuclear Medicine department for myocardial viability assessment
Sampling Method: Non-Probability Sample
Enrollment: 75
Dates: Start 2003-10; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Alain Manrique, MD, Study Chair — University Hospital, Rouen; Pierre-Yves Marie, MD, Study Director — Central Hospital, Nancy, France; Philippe Franken, MD, Study Director — Free University of Brussels
Locations (8):
- AZ-VUB, Brussels, Belgium
- France (7):
  - Hopital Avicenne, Bobigny
  - CHU de Brest, Brest
  - University Hospital of Caen, Caen
  - Hopital Sud-Francilien, Corbeil
  - University Hospital of Nancy, Nancy
  - Hopital Européen Georges Pompidou, Paris
  - University Hospital of Rouen, Rouen

REFERENCES:
- [Background] Allman KC, Shaw LJ, Hachamovitch R, Udelson JE. Myocardial viability testing and impact of revascularization on prognosis in patients with coronary artery disease and left ventricular dysfunction: a meta-analysis. J Am Coll Cardiol. 2002 Apr 3;39(7):1151-8. doi: 10.1016/s0735-1097(02)01726-6. PMID 11923039
- [Background] Everaert H, Vanhove C, Franken PR. Effects of low-dose dobutamine on left ventricular function in normal subjects as assessed by gated single-photon emission tomography myocardial perfusion studies. Eur J Nucl Med. 1999 Oct;26(10):1298-303. doi: 10.1007/s002590050586. PMID 10541828
- [Background] Everaert H, Vanhove C, Franken PR. Effect of beta-blockade on low-dose dobutamine-induced changes in left ventricular function in healthy volunteers: assessment by gated SPET myocardial perfusion scintigraphy. Eur J Nucl Med. 2000 Apr;27(4):419-24. doi: 10.1007/s002590050525. PMID 10805115
- [Background] Leoncini M, Sciagra R, Maioli M, Bellandi F, Marcucci G, Sestini S, Chiocchini S, Dabizzi RP. Usefulness of dobutamine Tc-99m sestamibi-gated single-photon emission computed tomography for prediction of left ventricular ejection fraction outcome after coronary revascularization for ischemic cardiomyopathy. Am J Cardiol. 2002 Apr 1;89(7):817-21. doi: 10.1016/s0002-9149(02)02203-8. PMID 11909565